CLINICAL TRIAL: NCT00390182
Title: GCC 0319: Low Dose Upper Abdominal Radiation Therapy (LD-UART) + Gemcitabine in Patients With Advanced, Unresectable Pancreatic Cancer (PC)
Brief Title: Low Dose Upper Abdominal Radiation Therapy (LD-UART) + Gemcitabine in Patients With Advanced, Unresectable Pancreatic Cancer (PC)
Acronym: GCC0319
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00042314
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Gastrointestinal Neoplasms; Ovarian Neoplasms
Keywords: GI tumors; Locally Advanced; Metastatic; Hepatobiliary; Ovary
MeSH Terms: conditions — Gastrointestinal Neoplasms; Ovarian Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Gemcitabine will be given at 1250 mg per meter squared over 2 hours days 1 and 8 of a 21 day cycle for a total of 4 cycles.
  Radiation: External Radiation Therapy The total dose would be 19.2 Gy divided over 32 fractions twice a day, on day 1 and day 8 after chemotherapy.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine will be given at 1250 mg per meter squared over 2 hours days 1 and 8 of a 21 day cycle for a total of 4 cycles.
  Radiation:External Radiation Therapy The total dose would be 19.2 Gy divided over 32 fractions twice a day, on day 1 and day 8 after chemotherapy.
  **Radiation is the experimental part of the study.
  Other Names: Gemzar; Radiation:External Radiation Therapy; **Radiation is the experimental part of the study.

SUMMARY:
The purposes of this study are:

1. To assess the maximum tolerated dose of low-dose UART(Upper Abdominal Radiation Therapy ) or WART(Whole Abdominal Radiation Therapy) given in combination with standard fixed dose-rate Gemcitabine in patients with advanced gastrointestinal (GI) or ovarian tumors (Phase I).
2. To assess response rate and survival in advanced upper GI tumors following completion of therapy (Phase II).

DETAILED DESCRIPTION:
Before entering this study the doctor will examine the patient and order blood tests. These tests will use approximately 10 ml of blood. Blood work should be done within 3 weeks prior to treatment.. Women of child-bearing potential are required to have a pregnancy test done within 7 days prior to the start of treatment . A CT or a PET/CT scan of the chest, abdomen and pelvis will be done within 4 weeks prior to starting treatment . All subjects participating in this study will receive radiation therapy and chemotherapy. Patients will get 4 cycles of chemotherapy along with radiation. Each cycle of chemotherapy consists of gemcitabine given i.v. on day 1 and day 8 of treatment. XRT is given on days 1 and 2 and on days 8 and 9 twice a day. This works out to 8 treatments of XRT per course of chemo. Overall, a total of 32 treatments of radiation therapy will be given during the 4 sessions of chemotherapy. Blood work for CBC with differential and platelets will be done prior to each dose of chemotherapy.The investigational portion of this study is the radiation therapy given to the abdomen on the same day and the day after the patient receives chemotherapy. Three-Four weeks after treatment completion the patient will be evaluated again. The treating physician will examine the patient and order blood tests. These tests will use approximately 10 ml of blood. The physician will also order a repeat CT or PET/CT to compare the disease status after treatment. These tests are not experimental and are part of routine check-ups of patients with pancreatic cancer. Patients will be followed for survival. Protected health information will not be reviewed by someone other than the patient's provider to identify potential subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are eligible if they have newly diagnosed histologically confirmed locally advanced or metastatic tumors of the pancreas. Patients must be felt to be unresectable by surgical criteria or felt to be medically inoperable. Patients may also be Stage IV with metastatic disease to the liver. Patients with bone and/or lung metastasis may be included at the investigators discretion.
2. Patients must have measurable disease by CT scan.
3. Patients must be able to give informed consent. Patients must be older than 18 years of age.
4. Patients should have adequate bone marrow, renal, and hepatic function including: Bilirubin less than 1.25 x institutional normal LDH SGPT, SGOT, and alkaline phosphatase less than3 x institutional normal Serum creatinine less than or equal to 3 mg/dl. Absolute neutrophil count of greater than 1500 Hemoglobin greater than 9 gm per dl Platelet count greater than 100,000 WBC greater than 3000 cells per mcl
5. Women of child-bearing potential must be agreeable to adequate contraception.(hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.)
6. Patients must have a Karnofsky performance status of greater than or equal 60 or Zubrod of less or equal to 2.
7. Life expectancy of at least 3 months.
8. May have had a second malignancy or multiple malignancies if adequately controlled by clinical means. patients with more than one type of cancer must be cleared by the principal investigator.
9. Patients must be at least 1 week from any major operative procedure.

10 .Patients may have brain metastasis if these brain metastasis are well controlled by usual clinical criteria and if the life expectancy is at least 3 months. Any patient with brain metastasis must be cleared by the principal investigator.

Exclusion Criteria:

1. Active infection requiring intravenous (IV) antibiotics at the time of entry.
2. Cerebral metastasis which has not been adequately controlled.
3. Significant malnutrition, cachexia, inundation or inability to give informed consent by clinical assessment.
4. Concurrent chemotherapy not prescribed in this protocol.
5. Any significant medical problems such as diabetes, cardiomyopathy or hypertension which is not reasonably controlled
6. Prior radiation or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Regine, MD, Principal Investigator — Chair - University of Maryland
Locations (2):
- University of Maryland & Baltimore VA medical centre, Baltimore, Maryland, United States
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients with cancer are seen by a multi-discipline clinic (medical, surgical, radiotherapy, etc). The PI or Co-PI identifies eligible candidates and initiates the discussion of research participation.
Groups:
- Gem(1250mg/m2, d1, 8) +LDFRT (60cGy/fx BID, d1,2,8,9): 4 cycles (1 cycle = 21 days): Gemcitabine 1250/m2 given IV Day 1 and Day 8; with concurrent Low Dose Fractionated Radiation Therapy (LDFRT). The total Radiation dose would be 19.2 Gy divided over 32 fractions. Treatment will be given in 2 fractions with a minimum 4 hr inter-fraction interval, not to exceed 6 hours. Radiotherapy given after the initiation of Gemcitabine Days 1,2,8, and 9.
Period: Overall Study
Arm/Group | Gem(1250mg/m2, d1, 8) +LDFRT (60cGy/fx BID, d1,2,8,9)
Started | 38
Completed | 33
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Standard Chemotherapy, Gemcitabine With Concurrent Low Dose Ra
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 29
  Canada | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 3 weeks
Measure: Number; unit: participants
Groups:
- Low Dose Fractionated Radiation Therapy (LDFRT) + Gemcitabine: Use of LDFRT with systemic gemcitabine is safe, tolerable, and potentially effective. In advanced pancreatic cancer, where response rates with single agent gemcitabine have been low, this chemopotentiation paradigm may improve survival among a poor prognostic patient cohort.
Arm/Group | Low Dose Fractionated Radiation Therapy (LDFRT) + Gemcitabine
Number analyzed (Participants) | 25
participants | 3 [2.7 to 23.1]

2. Other Pre Specified Outcome: Percentage of Participants With Distant Mestastases - Liver
Description: Patients with distant mestastases to the liver
Time Frame: Participants were followed for an average of 8 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Dose Fractionated Radiation Therapy (LDFRT) + Gemcitabine
Number analyzed (Participants) | 38
percentage of participants | 63 [45 to 78]

3. Other Pre Specified Outcome: Time of Advanced/Recurrent Disease Without Distant Metastases.
Description: Locally advanced/recurrent disease without distant metastases.
Time Frame: Participants were followed for an average of 8 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Low Dose Fractionated Radiation Therapy (LDFRT) + Gemcitabine
Number analyzed (Participants) | 16
months | 7.5 [5 to 13]

ADVERSE EVENTS:
Arm/Group | Standard Chemotherapy, Gemcitabine With Concurrent Low Dose Ra
Serious Adverse Events (participants affected / at risk) | 17/38
Other Adverse Events (participants affected / at risk) | 4/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Chemotherapy, Gemcitabine With Concurrent Low Dose Ra (N=38)
Hematologic (Blood and lymphatic system disorders) | 17 (25) — Hematologic toxicities, (combined any WBC, HGB, PLTs, ANC) grade 4 experienced in 17 out of 38 participants.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Chemotherapy, Gemcitabine With Concurrent Low Dose Ra (N=38)
Infection - non-neutropenic (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No